CLINICAL TRIAL: NCT01857843
Title: Early Effects of Intensive Lipid Lowering Treatment With Ezetimibe/ Simvastatin (Vytorin®) Assessed by Virtual Histology-Intravascular Ultrasound (VH-IVUS) and Optical Coherence Tomography (OCT) on Plaque Characteristics in Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2009-0032
Record Dates: First submitted 2013-05-15; First posted 2013-05-20 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ezetimibe; Simvastatin; Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ZES group (Experimental)
  Interventions: Device: Zotalolimus Eluting Stent
- EES group (Active Comparator)
  Interventions: Device: Everolimus eluting stent
- Vytorin group (Experimental)
  Interventions: Drug: Ezetimibe 10mg & Simvastatin 40mg
- Mevalotin group (Active Comparator)
  Interventions: Drug: Pravastatin 20mg

INTERVENTIONS:
Device: Zotalolimus Eluting Stent — Permuted block randomization into 4 groups according to the type of drug and stent will be carried out in a ratio of 1:1:1:1(i.e.,Vytorin-ZES, Vytorin-EES, mevalotin-ZES, or mevalotin-EES) for balanced randomization.
  Patients with native coronary arteries who fulfill all enrollment criteria for OCT study will be randomized to receive either ZES (Endeavor®-Sprint or Resolute-integrity) or EES (Xience®) in a ratio of 1:1.
  Arms: ZES group
Device: Everolimus eluting stent — Permuted block randomization into 4 groups according to the type of drug and stent will be carried out in a ratio of 1:1:1:1(i.e.,Vytorin-ZES, Vytorin-EES, mevalotin-ZES, or mevalotin-EES) for balanced randomization.
  Patients with native coronary arteries who fulfill all enrollment criteria for OCT study will be randomized to receive either ZES (Endeavor®-Sprint or resolute-integrity) or EES (Xience®) in a ratio of 1:1.
  Arms: EES group
Drug: Ezetimibe 10mg & Simvastatin 40mg — Permuted block randomization into 4 groups according to the type of drug and stent will be carried out in a ratio of 1:1:1:1(i.e.,Vytorin-ZES, Vytorin-EES, mevalotin-ZES, or mevalotin-EES) for balanced randomization.
  Patients will be randomized in a ratio of 1:1 according to the two different types of lipid lowering treatment.
  1. Ezetimibe 10mg/Simvastatin 40mg (Vytorin®, MSD)
  2. Pravastatin 20mg (mevalotin®, BMS)
  Arms: Vytorin group
Drug: Pravastatin 20mg — Permuted block randomization into 4 groups according to the type of drug and stent will be carried out in a ratio of 1:1:1:1(i.e.,Vytorin-ZES, Vytorin-EES, mevalotin-ZES, or mevalotin-EES) for balanced randomization.
  Patients will be randomized in a ratio of 1:1 according to the two different types of lipid lowering treatment.
  1. Ezetimibe 10mg/Simvastatin 40mg (Vytorin®, MSD)
  2. Pravastatin 20mg (mevalotin®, BMS)
  Arms: Mevalotin group

SUMMARY:
Objective: To evaluate the early effects of intensive lipid lowering treatments with ezetimibe/simvastatin (Vytorin®) for each component of coronary plaques.

Study Design

* Prospective, randomized, single-center study of each 80 subjects enrolled
* Subjects with acute coronary syndrome who meet all inclusion and exclusion criteria will be enrolled.
* Eligible subjects will be randomized 1:1 to A) Ezetimibe/Simvastatin (n=80) vs. B) Pravastatin (n=80), and each group of patients will be randomized further in a ratio of 1:1 to a) ZES (n=40) vs. b) EES (n=40), according to the type of stent used.
* All subjects will undergo VH-IVUS at initial procedure.
* Follow-up VH-IVUS will be performed at 3 months after index procedure. OCT at initial procedure and 3-months will be performed in available cases.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria

1. Acute coronary syndrome including unstable angina, acute non-ST elevation myocardial infarction and acute ST elevation myocardial infarction
2. Age of 20 years or older
3. Patients with signed informed consent

Angiographic inclusion criteria

1. De novo lesion without significant plaque (angiographic lumen diameter stenosis < 50%)
2. Reference vessel diameter ?> 3.0 mm by operator assessment
3. Segment length of 10-20 mm
4. Distance from the PCI site > 5.0mm (either proximal or distal)
5. Available for serial high quality IVUS studies of the entire segment.

Exclusion Criteria:

1. Failed PCI
2. Recommended coronary artery bypass grafting (CABG)
3. Cardiogenic Shock
4. Administration of lipid lowering agents before enrollment
5. Significant hepatic dysfunction (3 times normal reference values)
6. Significant renal dysfunction (Serum creatinine > 2.0 mg/dl)
7. Significant leukopenia, thrombocytopenia, anemia, or known bleeding diathesis
8. Pregnant women or women with potential childbearing
9. Saphenous vein graft

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-11; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Quantitative change in fibrofatty component of plaque measured by VH-IVUS | baseline and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea